CLINICAL TRIAL: NCT06642597
Title: An International, Multi-centre, Randomised Controlled Trial Co-designed With Consumers With Lived Experience of Peritoneal Dialysis (PD) to Determine the Optimal Approach to Starting Patients With Kidney Failure on PD
Brief Title: STarting incrEmental Prescription of Peritoneal Dialysis
Acronym: STEP-PD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Queensland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AKTN 24.01
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Peritoneal Dialysis (PD); Kidney Failure
Keywords: Kidney failure; Kidney disease; peritoneal dialysis; incremental start PD
MeSH Terms: conditions — Renal Insufficiency; Kidney Diseases

STUDY DESIGN:
Intervention Model Description: Multicentre, prospective, adaptive, randomised, open-label, parallel group, non-inferiority trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Incremental PD (Experimental): Incremental PD: Commence PD using goal-directed PD prescription ≤14 exchanges/week for continuous ambulatory PD (CAPD) or ≤21 exchanges/week for automated PD (APD) with no day dwell until an indication for increase in the PD dose (trigger point) is reached.
  Interventions: Other: Incremental PD
- Full dose PD (Active Comparator): Full dose PD: Commence with 24 hours, 7 days/week PD (i.e., CAPD ≥28 exchanges/week or APD (overnight) with day dwell (i.e., no dry abdomen)).
  Interventions: Other: Full dose PD

INTERVENTIONS:
Other: Incremental PD — Incremental PD: Commence PD using goal-directed PD prescription ≤14 exchanges/week for continuous ambulatory PD (CAPD) or ≤21 exchanges/week for automated PD (APD) with no day dwell until an indication for increase in the PD dose (trigger point) is reached.
  Arms: Incremental PD
Other: Full dose PD — Full dose PD: Commence with 24 hours, 7 days/week PD (i.e., CAPD ≥28 exchanges/week or APD (overnight) with day dwell (i.e., no dry abdomen)).
  Arms: Full dose PD

SUMMARY:
Kidney failure is fatal without dialysis. Peritoneal dialysis (PD) completed at home offers greater flexibility and autonomy for patients . However, PD is often prescribed for 24 hours/day, 7 days/week for every patient starting dialysis. This practice is not evidence-informed, may be unnecessary and potentially harmful. The STEP-PD trial aims to determine the optimal approach to commencing patients on PD through starting at low dose PD and incrementing over time.

DETAILED DESCRIPTION:
The STEP-PD study is an investigator-initiated, pragmatic, international, multicentre, prospective, adaptive, randomised, open-label, parallel group, non-inferiority trial led by an international multi-disciplinary team of clinician scientists, nephrologists, consumers, social scientists, trialists, health economists, dialysis nurses, statisticians, and registry experts. The STEP-PD trial is co-designed with consumers with lived experience of peritoneal dialysis (PD) to determine the optimal approach to starting patients with kidney failure on PD. Specifically, this trial will test the hypothesis that, compared with full dose PD, starting patients on incremental start PD preserves symptom burden related quality of life (QOL), reduces dialysis burden, is safe, is more environmentally sustainable and costs less for patients, the community and the healthcare system. The STEP-PD trial has the potential to transform and personalise the treatment of kidney failure globally by providing definitive evidence on the patient-prioritised question regarding the effectiveness and safety of incremental start PD, particularly in relation to the patient-critical outcome of symptom burden-related QOL. Favourable results would lead to a paradigm shift in how patients are started on PD, thereby mitigating unnecessarily burdensome, expensive, and possibly harmful treatment.

ELIGIBILITY:
Inclusion Criteria:

* adults (≥18 years) commencing PD as their first dialysis therapy (and been on dialysis for <1 month)
* able to give informed consent

Exclusion Criteria:

* urine output <0.5L/day
* previous kidney transplant
* unlikely to be on dialysis for ≥1 year.
* known or planned pregnancy during the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2025-09-19 (Actual); Primary Completion 2029-09-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Quality of Life (QoL) | From enrollment to the end of treatment at 6 months
  Symptom burden-related QOL 6 months after dialysis start, assessed by the Symptoms and Problems of Kidney Disease (SPKD) component of KDQOL-36 (0 to 100; worst to best).

SECONDARY OUTCOMES:
Residual Kidney Function (RKF) | From enrollment to 3, 6, 9, 12 and 18 months
  Slope of RKF decline over time modelled with linear regression of the arithmetic means of 24-hour urinary urea and creatinine clearances at months 3, 6, 9, 12 and 18
Anuria | From enrollment to 3, 6, 9, 12 and 18 months
  Proportion of patients with anuria (<100mL/24h) at months 3, 6, 9, 12 and 18
Serious adverse event | Enrollment to 18 months
  Number of category type of serious adverse events
Death | Enrollment to 18 months
  Time to all-cause mortality
Major cardiovascular event | Enrollment to 18 months
  Time to first major cardiovascular event (defined as acute myocardial infarction)
Peritonitis | Enrollment to 18 months
  Time to first peritonitis event
Non-elective hospitalisations | Enrollment to 18 months
  Number of non-elective hospital admissions
Hospitalisations | Enrollment to 18 months
  Hospitalisation for fluid overload, hyperkalaemia, or uraemic complications; episodes of hyperkalaemia (≥6mmol/L)
Quality of Life (QOL) and life participation | Enrollment to 18 months
  QOL and life participation: quarterly KDQOL-36 (physical and mental composite scores; effects and burden of kidney disease) and the SF6D (a component of the KDQOL)

CONTACTS AND LOCATIONS:
Locations (3):
- Australia (2):
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Eastern Health, Box Hill, Victoria
- Taichung Veterans General Hospital, Taichung, Xitun District, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Data sets will be made available to researchers within STEP-PD for analysis of sub-studies and country-specific outcomes after the primary manuscript has been accepted for publication.
  For researchers outside STEP-PD, individual participant data will be made available upon request to a Data Access Committee, a review board set up to assess proposals based on sound science, benefit-risk balancing, and research team expertise. Ethics approval will be required. This process will be in effect for a period of 2 to 5 years following publication of the main study results.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: A period of 2 to 5 years following publication of the main study results.